CLINICAL TRIAL: NCT00112346
Title: A Randomized Multicenter Phase II Study of Gemcitabine/Platinum/Cetuximab Versus Gemcitabine/Platinum as First-Line Treatment for Patients With Advanced/Metastatic Non-Small Cell Lung Cancer
Brief Title: Study of Gemcitabine/Platinum +/- Cetuximab as First-Line Treatment for Patients With Advanced/Metastatic Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA225-100
Record Dates: First submitted 2005-06-01; First posted 2005-06-02 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Non-Small-Cell Lung Carcinoma
Keywords: Non-Small Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cetuximab; Platinum; Gemcitabine

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Cetuximab + platinum + gemcitabine
- B (Active Comparator)
  Interventions: Drug: Platinum + Gemcitabine

INTERVENTIONS:
Drug: Cetuximab + platinum + gemcitabine — Solution, IV, Cetuximab: 400mg/m2 on Day 1 then given weekly at 250mg/m2 starting on Day 8 + Gemcitabine given at 1250mg/m2 (Day 1 & Day 8 of each cycle) + Cisplatin given at 75mg/m2 or Carboplatin AUC=5, Cycle of therapy is every 3 weeks. Cetuximab is given weekly, Maximum of 6 cycles (18 weeks) Cetuximab will be continued during the period following discontinuation of chemotherapy, until disease progression or cetuximab intolerance.
  Other Names: Erbitux
  Arms: A
Drug: Platinum + Gemcitabine — Solution, IV, Gemcitabine given at 1250mg/m2 (Day 1 & Day 8 of each cycle) + Cisplatin given at 75mg/m2 or Carboplatin AUC=5, Cycle of therapy is every 3 weeks, Maximum of 6 cycles = 18 weeks.
  Arms: B

SUMMARY:
The primary purpose of this study is to estimate the number of patients with non-small cell lung cancer whose tumor responds to the treatments given in this study.

ELIGIBILITY:
Inclusion Criteria:

* Must have advanced or metastatic non-small cell lung cancer that has not been previously treated with any chemotherapy.
* Must not have received cetuximab or any medications that target the same pathway as cetuximab (such as Iressa or Tarceva).
* Must not have had hypersensitivity or severe allergic reactions to any monoclonal antibodies and must not have severe restrictive or interstitial lung disease.
* Must be able to carry out work of light or sedentary nature (e.g. light house work, office work).
* It must be at least 4 weeks since last major surgery or prior treatment with an investigational product and at least 12 weeks from any radiation therapy to the chest.

Exclusion Criteria:

* Women who are pregnant or breastfeeding.
* Women with a positive pregnancy test on enrollment or prior to study drug administration.
* Any concurrent malignancy (subjects with a previous malignancy but without evidence of disease for 5 years will be allowed to enter the trial).
* Symptomatic or uncontrolled metastases in the central nervous system (CNS).
* Peripheral neuropathy.
* Inadequate hematologic function defined by an absolute neutrophil count (ANC) <1,500/mm^3, a platelet count <100,000/mm^3, or a hemoglobin level < 9g/dL.
* Inadequate liver function.
* Inadequate kidney function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2005-01; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
tumor response per treatment arm

SECONDARY OUTCOMES:
disease control, symptom response, symptomatic progression, & progression free survival.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (38):
- United States (31):
  - Local Institution, Mobile, Alabama
  - Local Institution, Anchorage, Alaska
  - Local Institution, Bakersfield, California
  - Local Institution, Corona, California
  - Local Institution, Oxnard, California
  - Local Institution, San Diego, California
  - Local Institution, Whittier, California
  - Local Institution, Lakewood, Colorado
  - Local Institution, Boynton Beach, Florida
  - Local Institution, Brooksville, Florida
  - Local Institution, Inverness, Florida
  - Local Institution, Pembroke Pines, Florida
  - Local Institution, Austell, Georgia
  - Local Institution, Honolulu, Hawaii
  - Local Institution, Skokie, Illinois
  - Local Institution, Muncie, Indiana
  - Local Institution, Annapolis, Maryland
  - Local Institution, Frederick, Maryland
  - Local Institution, Rockville, Maryland
  - Local Institution, Plymouth, Massachusetts
  - Local Institution, Farmington, New Mexico
  - Local Institution, Armonk, New York
  - Local Institution, Stony Brook, New York
  - Local Institution, Gastonia, North Carolina
  - Local Institution, Wilmington, North Carolina
  - Local Institution, Bismarck, North Dakota
  - Local Institution, Cincinnati, Ohio
  - Local Institution, Portland, Oregon
  - Local Institution, Charleston, South Carolina
  - Local Institution, Dallas, Texas
  - Local Institution, Vancouver, Washington
- Canada (7):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Moncton, New Brunswick
  - Local Institution, Hamilton, Ontario
  - Local Institution, Montreal, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Windsor, Ontario
  - Local Institution, Greenfield Park, Quebec